CLINICAL TRIAL: NCT04135352
Title: A Phase 1/1b, Open-label Clinical Study of Intratumoral/Intralesional Administration of V938 in Combination With Pembrolizumab (MK-3475) in Participants With Advanced/Metastatic or Recurrent Malignancies
Brief Title: A Study of Intratumoral/Intralesional Administration of V938 in Combination With Pembrolizumab (MK-3475) in Participants With Advanced/Metastatic or Recurrent Malignancies (V938-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: V938-001; V938-001 (Other: MSD Protocol Number); 2020-003431-25 (EudraCT Number)
Record Dates: First submitted 2019-10-10; First posted 2019-10-22 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Neoplasm Metastasis
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Neoplasm Metastasis; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- V938 Dose A + delayed pembrolizumab (Experimental): This arm will enroll participants with advanced/metastatic or recurrent solid tumors. Participants receive Dose A of V938 intratumorally in cycles 1-7. Participants also receive 200 mg of pembrolizumab intravenously once every 3 weeks (Q3W) beginning with cycle 2 for a maximum of 35 cycles. Each cycle is 21 days.
  Interventions: Drug: 200 mg of pembrolizumab; Biological: V938
- V938 Dose B + delayed pembrolizumab (Experimental): This arm will enroll participants with advanced/metastatic or recurrent solid tumors. Participants receive Dose B of V938 intratumorally in cycles 1-7. Participants also receive 200 mg of pembrolizumab intravenously Q3W beginning with cycle 2 for a maximum of 35 cycles. Each cycle is 21 days.
  Interventions: Drug: 200 mg of pembrolizumab; Biological: V938
- V938 Dose C + delayed pembrolizumab (Experimental): This arm will enroll participants with advanced/metastatic or recurrent solid tumors. Participants receive Dose C of V938 intratumorally in cycles 1-7. Participants also receive 200 mg of pembrolizumab intravenously Q3W beginning with cycle 2 for a maximum of 35 cycles. Each cycle is 21 days.
  Interventions: Drug: 200 mg of pembrolizumab; Biological: V938
- V938 Dose D + delayed pembrolizumab (Experimental): This arm will enroll participants with advanced/metastatic or recurrent solid tumors. Participants receive Dose D of V938 intratumorally in cycles 1-7. Participants also receive 200 mg of pembrolizumab intravenously Q3W beginning with cycle 2 for a maximum of 35 cycles. Each cycle is 21 days.
  Interventions: Drug: 200 mg of pembrolizumab; Biological: V938
- V938 Dose B + immediate pembrolizumab (Experimental): This arm will enroll participants with advanced/metastatic or recurrent solid tumors. Participants receive Dose B of V938 intratumorally in cycles 1-7. Participants also receive 200 mg of pembrolizumab intravenously Q3W beginning with cycle 1 for a maximum of 35 cycles. Each cycle is 21 days.
  Interventions: Drug: 200 mg of pembrolizumab; Biological: V938
- V938 Dose C + immediate pembrolizumab (Experimental): This arm will enroll participants with advanced/metastatic or recurrent solid tumors. Participants receive Dose C of V938 intratumorally in cycles 1-7. Participants also receive 200 mg of pembrolizumab intravenously Q3W beginning with cycle 1 for a maximum of 35 cycles. Each cycle is 21 days.
  Interventions: Drug: 200 mg of pembrolizumab; Biological: V938
- V938 Dose D + immediate pembrolizumab (Experimental): This arm will enroll participants with advanced/metastatic or recurrent solid tumors. Participants receive Dose D of V938 intratumorally in cycles 1-7. Participants also receive 200 mg of pembrolizumab intravenously Q3W beginning with cycle 1 for a maximum of 35 cycles. Each cycle is 21 days.
  Interventions: Drug: 200 mg of pembrolizumab; Biological: V938
- Dose Expansion Arm A, Melanoma (Experimental): This arm will enroll only participants with with a diagnosis of stage III (unresectable) and Stage IV melanoma (any line of therapy). Participants receive V938 at the recommended Phase 2 Dose, determined by analysis of the Dose A-C arms, intratumorally in cycles 1-7. Participants also receive 200 mg of pembrolizumab intravenously Q3W beginning with cycle 1 for a maximum of 35 cycles. Each cycle is 21 days.
  Interventions: Drug: 200 mg of pembrolizumab; Biological: V938
- Dose Expansion Arm B, HNSCC (Experimental): This arm will only enroll participants with a diagnosis of advanced/metastatic head and neck squamous cell carcinoma (HNSCC). Participants receive V938 at the recommended Phase 2 Dose, determined by analysis of the Dose A-C arms, intratumorally in cycles 1-7. Participants also receive 200 mg of pembrolizumab intravenously Q3W beginning with cycle 1 for a maximum of 35 cycles. Each cycle is 21 days.
  Interventions: Drug: 200 mg of pembrolizumab; Biological: V938

INTERVENTIONS:
Drug: 200 mg of pembrolizumab — Participants receive 200 mg of pembrolizumab intravenously Q3W for a maximum of 35 21-day cycles.
  Other Names: MK-3475
Biological: V938 — Participants receive V938 intratumorally in cycles 1-7. Each cycle is 21 days.

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, pharmacokinetics, and V938 shedding in participants with advanced/metastatic or recurrent malignancies who receive V938 in combination with pembrolizumab (MK-3475). The primary objective is to determine the safety and tolerability and to identify a recommended Phase 2 dose (RP2D) of V938 administered in combination with pembrolizumab.

DETAILED DESCRIPTION:
Due to discontinuation of V938-001, all ongoing participants who completed V938 plus pembrolizumab treatment may be enrolled in an extension study (KN587) to continue pembrolizumab monotherapy for a total of 35 cycles since the first dose in V938-001 and to be monitored as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* For Dose-escalation arms (Doses A-D): Have a histologically confirmed advanced/metastatic solid tumor and have received, been intolerant to, or been ineligible for treatments known to confer clinical benefit.
* For Dose Expansion Arm A: Have a histologically confirmed Stage III (unresectable) or Stage IV cutaneous melanoma and have received and progressed following 1 or 2 prior lines of systemic treatments for metastatic melanoma which must include 1 line of treatment with PD-1 or PD-L1 immune checkpoint inhibitor either as monotherapy or in combination with other therapy.
* For Dose Expansion Arm B: Have a histologically confirmed advanced head and neck squamous cell carcinoma (HNSCC) and have received and progressed following 1 or 2 prior lines of systemic treatments for metastatic HNSCC which must include 1 line of treatment with PD-1 or PD-L1 immune checkpoint inhibitor either as monotherapy or in combination with other therapy.
* For Dose Expansion Arms A and B: Have at least 1 lesion that is amenable to both intratumoral (IT) injection and biopsy and have at least 1 distant and/or discrete noninjected lesion that is measurable per RECIST 1.1 criteria.
* For Dose-escalation Cohorts 2a, 3a, or 4a and Expansion Cohorts (Arms A and B) ONLY: Have baseline biopsy performed from 1 of the injectable lesions that are planned for IT injection and with tumor tissue provided.
* For all arms: Have at least 1 cutaneous or subcutaneous lesion amenable to IT injection and must be measurable and meet 1 of the following criteria per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1):

  * A cutaneous or subcutaneous lesion ≥1 cm in longest diameter for solid tumors, or ≥1.5 cm in short axis for a nodal lesion in participants with solid tumor. The longest diameter for an injectable lesion must be ≤10 cm for both solid tumors and nodal lesions in participants with solid tumors.
  * Multiple coalescing, superficial lesions that in aggregate have a longest diameter of ≥1 cm and ≤10 cm.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Show adequate organ function.
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 120 days: either be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent, OR must agree to use contraception unless confirmed to be azoospermic. Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP)
  * Is a WOCBP and using a contraceptive method that is highly effective, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 120 days after the last dose of study intervention.
* HIV-infected participants must have well controlled HIV on antiretroviral therapy (ART), per study criteria.

Exclusion Criteria:

* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) prior to the first dose of study intervention or has not recovered from any adverse events (AEs) that were due to cancer therapeutics administered more than 4 weeks earlier. Participants receiving ongoing replacement hormone therapy for endocrine immune-related AEs will not be excluded from participation in this study.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer or in situ cervical cancer, or other in-situ cancers.
* Has clinically active central nervous system metastases and/or carcinomatous meningitis.
* Has had a severe hypersensitivity reaction to treatment with the monoclonal antibody/components of the study intervention or has a history of any contraindication or has a severe hypersensitivity to any components of pembrolizumab (≥Grade 3).
* Has an active infection requiring therapy.
* Has a history of (noninfectious) pneumonitis that required steroids or current pneumonitis.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years except vitiligo or resolved childhood asthma/atopy.
* Is on chronic systemic steroid therapy in excess of replacement doses (prednisone ≤10 mg/day is acceptable), or on any other form of immunosuppressive medication.
* Participants with known Hepatitis B or C infections or known to be positive for hepatitis B antigen/hepatitis B virus DNA or hepatitis C antibody or RNA.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study intervention.
* Has not fully recovered from any effects of major surgery without significant detectable infection.
* Has received a live-virus vaccine within 30 days of planned treatment start.
* Is currently participating and receiving study intervention in a study of an investigational agent or has participated and received study intervention in a study of an investigational agent or has used an investigational device within 28 days of administration of V938.
* Has a history of re-irradiation for HNSCC at the projected injection site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- United States (3):
  - UCSF Helen Diller Family Comprehensive Cancer Center ( Site 0002), San Francisco, California
  - MD Anderson Cancer Center ( Site 0001), Houston, Texas
  - Huntsman Cancer Institute ( Site 0004), Salt Lake City, Utah
- Princess Margaret Cancer Centre ( Site 0010), Toronto, Ontario, Canada
- Israel (2):
  - Rambam Health Care Campus-Oncology Division ( Site 0020), Haifa
  - Chaim Sheba Medical Center ( Site 0021), Ramat Gan

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants with advanced/metastatic or recurrent solid tumors.
Pre-assignment Details: The study was designed/ planned to have two parts: dose escalation and expansion cohorts. Due to termination of the study, dose expansion Arm A and Arm B were not started in the study.
Groups:
- Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab: This arm enrolled participants with advanced/metastatic or recurrent solid tumors. Participants received once every 3 weeks (Q3W) dose of 1x10^7 PFU of V938 intratumorally on day 1 (D1) in cycles 1-7. Participants also received 200 mg of pembrolizumab intravenously Q3W beginning with cycle 2 for a maximum of 35 cycles. Each cycle was 21 days.
- Cohort 2: V938 1x10^8 PFU + Pembrolizumab: This arm enrolled participants with advanced/metastatic or recurrent solid tumors. Participants received once Q3W dose of 1x10^8 PFU of V938 intratumorally on D1 in cycles 1-7. Participants also received 200 mg of pembrolizumab intravenously Q3W beginning with cycle 2 for a maximum of 35 cycles. Each cycle was 21 days.
- Cohort 3: V938 3x10^8 PFU + Pembrolizumab: This arm enrolled participants with advanced/metastatic or recurrent solid tumors. Participants received once Q3W dose of 3x10^8 of V938 intratumorally on D1 in cycles 1-7. Participants also received 200 mg of pembrolizumab intravenously Q3W beginning with cycle 2 for a maximum of 35 cycles. Each cycle was 21 days.
- Cohort 4: V938 5x10^8 PFU + Pembrolizumab: This arm enrolled participants with advanced/metastatic or recurrent solid tumors. Participants received once Q3W dose of 5x10^8 PFU of V938 intratumorally on D1 in cycles 1-7. Participants also received 200 mg of pembrolizumab intravenously Q3W beginning with cycle 2 for a maximum of 35 cycles. Each cycle was 21 days.
- Cohort 3a: V938 3x10^8 PFU + Pembrolizumab: This arm enrolled participants with advanced/metastatic or recurrent solid tumors. Participants received once Q3W dose of 3x10^8 PFU of V938 on D1 intratumorally in cycles 1-7. Participants also received 200 mg of pembrolizumab intravenously Q3W beginning with cycle 1 for a maximum of 35 cycles. Each cycle was 21 days.
- Cohort 4a: V938 5x10^8 PFU + Pembrolizumab: This arm enrolled participants with advanced/metastatic or recurrent solid tumors. Participants received once Q3W dose of 5x10^8 PFU of V938 intratumorally on D1 in cycles 1-7. Participants also received 200 mg of pembrolizumab intravenously Q3W beginning with cycle 1 for a maximum of 35 cycles. Each cycle was 21 days.
- Dose Expansion Arm A, Melanoma: This arm was intended enroll participants with diagnosis of stage III (unresectable) and Stage IV melanoma (any line of therapy). Participants were intended to receive V938 at the recommended Phase 2 dose, determined by analysis of the dose 1x10^7 PFU to 3x10^8 PFU arms, intratumorally on D1 in cycles 1-7. Participants were also intended to receive 200 mg of pembrolizumab intravenously Q3W beginning with cycle 1 for a maximum of 35 cycles. Each cycle was 21 days. Due to study termination, this arm was not started in the study.
- Dose Expansion Arm B, HNSCC: This arm was intended to enroll participants with a diagnosis of advanced/metastatic head and neck squamous cell carcinoma (HNSCC). Participants were intended to receive V938 at the recommended Phase 2 dose, determined by analysis of the dose 1x10^7 PFU to 3x10^8 PFU arms, intratumorally in cycles 1-7. Participants were also intended to receive 200 mg of pembrolizumab intravenously Q3W beginning with cycle 1 for a maximum of 35 cycles. Each cycle was 21 days. Due to study termination, this arm was not started in the study.
Period: Overall Study
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC
Started | 3 | 4 | 13 | 5 | 5 | 5 | 0 | 0
Treated | 3 | 4 | 12 (1 participant randomized in error and was not treated) | 5 | 5 | 5 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 13 | 5 | 5 | 5 | 0 | 0
Not completed — Not treated-randomization error | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 2 | 5 | 1 | 4 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 3 | 4 | 7 | 0 | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all participants who received received at least 1 dose of study intervention. Due to termination of the study, dose expansion Arm A and Arm B were not started in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC | Total
Number analyzed (Participants) | 3 | 4 | 13 | 5 | 5 | 5 | 0 | 0 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.3 (5.1) | 55.3 (4.2) | 60.3 (10.9) | 53.2 (13.0) | 67.8 (11.7) | 67.6 (9.2) |  |  | 61.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 6 | 4 | 1 | 3 | 0 | 0 | 17
  Male | 0 | 4 | 7 | 1 | 4 | 2 | 0 | 0 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 3 | 4 | 12 | 3 | 5 | 5 | 0 | 0 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 4 | 13 | 4 | 5 | 5 | 0 | 0 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature). The analysis population consisted of all participants who received received at least 1 dose of study intervention. Due to program prioritization, the study was terminated early in dose escalation. Due to termination of the study, dose expansion Arm A and Arm B were not started in the study.
  Participants
    ECOG = 0 | 2 | 0 | 6 | 2 | 2 | 2 | 0 | 0 | 14
    ECOG = 1 | 1 | 4 | 7 | 3 | 3 | 3 | 0 | 0 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicity (DLT)
Description: DLT was defined as a treatment-related adverse event (AE) including the following: Grade (Gr) 4 nonhematologic toxicity (not laboratory), Gr 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia or Gr 4 thrombocytopenia of any duration or Gr 3 thrombocytopenia associated with clinically significant bleeding, Gr 3 non-hematological AE with the exception of fatigue lasting ≤72 hours, Gr 3 nausea, vomiting, diarrhea or rash, any Gr 3 or Gr 4 nonhematologic that lead to hospitalization or abnormality persisting for >1 week or resulting in a drug induced liver injury (DILI), febrile neutropenia Gr 3 or Gr, prolonged delay (>2 weeks) in initiating cycle 3 (for Cohorts 1-4) or cycle 2 (for cohorts 2a-4a) due to study intervention-related toxicity, intervention-related toxicity that caused study discontinuation or missing >1 injection of V938 as a result of drug-related AE(s) during the first 2 cycles (for cohorts 1-4) or during the first cycle (for cohort 2a-4a), Gr 5 toxicity
Time Frame: Up to ~ 42 days for cohort 1, 2, 3 and 4; Up to ~ 21 days for cohorts 3a and 4a
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study intervention and who met the criteria for DLT evaluability. Due to termination of the study, dose expansion Arm A and Arm B were not started in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC
Number analyzed (Participants) | 3 | 4 | 11 | 5 | 5 | 5 | 0 | 0
Participants | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: Number of participants who experienced an AE defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study treatment
Time Frame: Up to ~ 28 months
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study intervention. Due to termination of the study, dose expansion Arm A and Arm B were not started in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC
Number analyzed (Participants) | 3 | 4 | 12 | 5 | 5 | 5 | 0 | 0
Participants | 2 | 4 | 12 | 5 | 5 | 5 | 0 | 0

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued treatment due to an AE was assessed.
Time Frame: Up to ~ 25 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC
Number analyzed (Participants) | 3 | 4 | 12 | 5 | 5 | 5 | 0 | 0
Participants | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions), as assessed by the investigator. In solid tumors, assessment will be based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) and modified RECIST 1.1 for immune-based therapeutics (iRECIST). The percentage of participants who experience a CR or PR based on the above criteria will be presented.
Time Frame: Up to ~ 33 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC
Number analyzed (Participants) | 3 | 4 | 12 | 5 | 5 | 5 | 0 | 0
Percentage of Participants | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 52.2] | 40.0 [5.3 to 85.3] |  |

5. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to 6 Hours Postdose (AUC0-6) for V938 Ribonucleic Acid (RNA) in Plasma
Description: The AUC0-6 for V938 RNA in plasma was calculated.
Time Frame: Cycle 1 (C1) Day1 (D1), C1D8 and C2D1. Each Cycle is 21 days.
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study intervention. Per protocol, AUC0-6 was calculated for the participants who had concentration values. Due to termination of the study, data were not collected for participants in Cohort 4a Cohort 4a: V938 5x10^8 PFU + pembrolizumab and dose expansion Arm A and Arm B were not started in the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*pfu/mL
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC
Number analyzed (Participants) | 3 | 4 | 12 | 5 | 5 | 0 | 0 | 0
Hours*pfu/mL
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 3 | 6 | 1 | 2 | 0 | 0 | 0
  Cycle 1 Day 1 | 1249 (157.1) | 55.5 (1007.4) | 354 (313.1) | 2520 (NA) — Coefficient of variation (CoV) not calculable due to n=1 | 430 (79.5) |  |  |
  Cycle 1 Day 8: number analyzed (Participants) | 1 | 3 | 8 | 1 | 3 | 0 | 0 | 0
  Cycle 1 Day 8 | 753 (NA) — CoV not calculable due to n=1 | 314 (307.1) | 191 (104.3) | 1040 (NA) — CoV not calculable due to n=1 | 95.7 (107.1) |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 5 | 1 | 2 | 0 | 0 | 0
  Cycle 2 Day 1 | 46.2 (14.6) | 158 (64.7) | 119 (239.8) | 867 (NA) — CoV not calculable due to n=1 | 24.4 (3.9) |  |  |

6. Secondary Outcome: Maximum Concentration (Cmax) of V938 Ribonucleic Acid (RNA) in Plasma
Description: The Cmax for V938 RNA in plasma was reported.
Time Frame: Cycle 1 (C1) Day1 (D1), C1D8 and C2D1. Each Cycle is 21 days.
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study intervention. Per protocol, Cmax was calculated for the participants who had concentration values. Due to termination of the study, data were not collected for participants in Cohort 4a Cohort 4a: V938 5x10^8 PFU + pembrolizumab and dose expansion Arm A and Arm B were not started in the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pfu/mL
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC
Number analyzed (Participants) | 3 | 4 | 12 | 5 | 5 | 0 | 0 | 0
pfu/mL
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 3 | 6 | 1 | 2 | 0 | 0 | 0
  Cycle 1 Day 1 | 65.6 (104.7) | 15.1 (951.6) | 55.6 (593.8) | 595 (NA) — CoV not calculable due to n=1 | 26.6 (3122.3) |  |  |
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 3 | 8 | 2 | 3 | 0 | 0 | 0
  Cycle 1 Day 8 | 66.4 (291.2) | 85.5 (176.0) | 57.6 (78.5) | 235 (17.7) | 10.1 (1259.0) |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 5 | 1 | 2 | 0 | 0 | 0
  Cycle 2 Day 1 | 11.2 (14.4) | 51.3 (77.4) | 31.0 (255.9) | 97.9 (204.1) | 8.40 (37.9) |  |  |

7. Secondary Outcome: Number of Participants With Newcastle Disease Virus (NDV) RNA Shedding Per Polymerase Chain Reaction (PCR)
Description: Shedding raises the possibility of transmission of oncolytic products from treated to untreated individuals. Participants treated with V938 may excrete virus via urine, respiratory tract, or GI tract after the V938 administration. The samples from the participants were collected for evaluation of virus shedding. The presence of V938 viral RNA (pfu/ml) using qRT-PCR assay was assessed in oral cavity/throat, urine, injection site, and anus to detrmine the environmental viral shedding.
Time Frame: Predose cycle 1 on 3 separate days, and cycles 3, 5, 8, 9, and 10 on day 1. 2 and 4-6 hours postdose cycle 1 day 1. Each cycle is 21 days.
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study intervention and had available data. Per protocol, V938 excretion was calculated for the participants who had concentration values. Due to termination of the study, dose expansion Arm A and Arm B were not started in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC
Number analyzed (Participants) | 3 | 4 | 11 | 5 | 5 | 5 | 0 | 0
Participants
  Oral cavity/throat: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Oral cavity/throat | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Urine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Injection site: number analyzed (Participants) | 3 | 4 | 10 | 0 | 0 | 0 | 0 | 0
  Injection site | 3 | 4 | 10 | 0 | 0 | 0 | 0 | 0
  Anal swab: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anal swab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With NDV Infectivity in Excretory Tissue Samples
Description: Participants treated with V938 may excrete virus via urine, respiratory tract, or GI tract after the V938 administration. The positive virus shedding samples that were analyzed in viral shedding were further assessed for NDV infectivity. NDV infectivity was measured by cell-based assay.
Time Frame: as for outcome 7
Population: The analysis population consisted of all randomized participants who received at least 1 dose of study intervention and had available data. V938 excretion based on infectivity was calculated for the participants who had concentration values. Due to termination of the study, dose expansion Arm A and Arm B were not started in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC
Number analyzed (Participants) | 3 | 4 | 12 | 5 | 5 | 5 | 0 | 0
Participants
  Oral cavity/throat: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Oral cavity/throat | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Injection site | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anal swab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to ~ 28 months
Description: All-cause mortality includes all allocated participants. AEs include participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE, unless related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment were excluded as AEs.
Arm/Group | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab | Cohort 2: V938 1x10^8 PFU + Pembrolizumab | Cohort 3: V938 3x10^8 PFU + Pembrolizumab | Cohort 4: V938 5x10^8 PFU + Pembrolizumab | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab | Dose Expansion Arm A, Melanoma | Dose Expansion Arm B, HNSCC
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/4 | 8/13 | 0/5 | 3/5 | 1/5 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/4 | 2/12 | 1/5 | 2/5 | 4/5 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/3 | 4/4 | 12/12 | 5/5 | 5/5 | 5/5 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab (N=3) | Cohort 2: V938 1x10^8 PFU + Pembrolizumab (N=4) | Cohort 3: V938 3x10^8 PFU + Pembrolizumab (N=12) | Cohort 4: V938 5x10^8 PFU + Pembrolizumab (N=5) | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab (N=5) | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab (N=5) | Dose Expansion Arm A, Melanoma (N=0) | Dose Expansion Arm B, HNSCC (N=0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Distributive shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: V938 1x10^7 Plaque-forming Units (PFU) + Pembrolizumab (N=3) | Cohort 2: V938 1x10^8 PFU + Pembrolizumab (N=4) | Cohort 3: V938 3x10^8 PFU + Pembrolizumab (N=12) | Cohort 4: V938 5x10^8 PFU + Pembrolizumab (N=5) | Cohort 3a: V938 3x10^8 PFU + Pembrolizumab (N=5) | Cohort 4a: V938 5x10^8 PFU + Pembrolizumab (N=5) | Dose Expansion Arm A, Melanoma (N=0) | Dose Expansion Arm B, HNSCC (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (9) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (2) | 2 (4) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (4) | 7 (10) | 4 (10) | 2 (3) | 5 (5) | 0 (0) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation mucositis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cortisol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Magnetic resonance imaging head abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Quadrantanopia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulite (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 3 (4) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Poor peripheral circulation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT04135352/Prot_SAP_000.pdf